CLINICAL TRIAL: NCT01803984
Title: MIBRAIN - Migraine and the Brain: Consequences, Causes, and Vascular Interaction
Acronym: MIBRAIN
Status: Terminated | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2012/19
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Migraine
Keywords: Migraine; Brain structure; MRI
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient with migraine with aura: Patients with a clearly defined migraine (as per IHS criteria) with aura, who are aged 30 and older and are able to fluently speak French.
  Interventions: Device: MRI; Device: EndoPAT; Other: Neuropsychological battery
- Patient with migraine without aura: patients with a clearly defined migraine (as per IHS criteria) without aura who are aged 30 and older, are able to fluently speak French, and who are willing to participate
  Interventions: Device: MRI; Device: EndoPAT; Other: Neuropsychological battery

INTERVENTIONS:
Device: MRI
Device: EndoPAT — The endothelial function will be measured with a noninvasive Peripheral Arterial Tone (PAT) signal technology using the EndoPAT device
Other: Neuropsychological battery — The cognitive status in the patient cohort will be ascertained by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS).

SUMMARY:
Migraine is a very common, chronic/intermittent and disabling neurovascular headache disorder that has long believed to have no severe consequences. Recent evidence, however, strongly suggest that migraine is associated with increased risk of ischemic stroke and there is initial evidence that migraine is associated with structural brain changes independent of the occurrence of stroke.

As migraine has strong links with the vascular system, it is plausible that vascular functions interact on the association between migraine and structural brain changes as well as cognition.

Our primary objectives are to investigate: (i) the relationship of migraine and migraine subtypes on magnetic resonance imaging (MRI) changes in a cohort of patients with active migraine; (ii) the relationship of migraine on cognitive performance among patients with active migraine; and (iii) the relationship of migraine and migraine specifics with vascular functions and morbidity. As secondary objective, we investigate whether the association of migraine on structural brain changes or cognitive performance is modified by vascular functions.

This will be an observational study conducted in the Headache Center in Bordeaux. 300 patients have to be included (150 patients with migraine with aura and 150 patients with migraine without aura).

Inclusion criteria are: all patients with a clearly defined migraine (as per IHS[International Headache Classification] criteria) who are aged 30 and older, are able to fluently speak French, and who are willing to participate.

Exclusion criteria are: pregnant woman and patient who have a major psychiatric disease or major anxiety disorder or had a pacemaker (which would not allow to perform a MRI imaging).

The cognitive status in the patient cohort will be ascertained by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). In addition to the RBANS, we will use the HIT-6 (Headache Impact Test) and MIDAS (MIgraine Disability ASessment) and the depression scale CES-D (Center for Epidemiologic Studies Depression Scale).

Vascular risk status will be assessed by measurement of blood pressure and reports of vascular risk factors. The endothelial function will be measured with a noninvasive Peripheral Arterial Tone (PAT) signal technology using the EndoPAT device (Itamar Medical Inc, Framingham, MA).

For crude comparisons, chi-square tests will be used for categorical variables and t-test for continuous variables. Multivariable-multinominal modeling techniques will be utilized for the comparisons adjusting for potential confounding variables. All statistical tests will be two-tailed and a P <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patient with migraine according to the criteria defined by the International Headache Society (ICHD-II)
* Patient aged 30 years old and older
* Patient speaking fluent french

Exclusion Criteria:

* pregnant woman
* patient with a serious psychiatric psychological illness
* patient having a serious anxiety (claustrophobia)
* Patient bearing an electronic or a metallic device (pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a clearly defined migraine (as per IHS criteria) who are aged 30 and older, are able to fluently speak French, do not have a major psychiatric disease or major anxiety disorder which would not allow to perform a MRI imaging, and who are willing to participate.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2013-03-22 (Actual); Primary Completion 2014-12-03 (Actual); Study Completion 2014-12-03 (Actual)

PRIMARY OUTCOMES:
Differences in magnetic resonance imaging (MRI) between migraine without aura and migraine with aura patients (frequency of hyperintensities, white matter lesions....) | Within 3 months after inclusion
Differences in the Total Score of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) between migraine without aura and migraine with aura patients. | Baseline
  The Total Score of the RBANS reflects the neurocognitive status of the patient by summing five index/domain scores. The domains are Immediate Memory, Visuospatial/Constructional, Language, Attention, and Delayed Memory.
Differences in the Reactive Hyperemia Index (RHI) and the Augmentation Index (AI) between migraine without aura and migraine with aura patients | Baseline
  RHI will measured by the non invasive endothelial peripheral arterial tomography (EndoPat 2000 Itamar Medical Ltd) device.

SECONDARY OUTCOMES:
Correlation between MRI and Total Score of RBANS with RHI / AI (endothelial function) between migraine groups. | Within 3 months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Tobias KURTH, MD, Principal Investigator — Inserm Unit 708 - Neuroépidemiologie
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, France